CLINICAL TRIAL: NCT00923013
Title: Randomized Trial of Cladribine (CdA) With Simultaneous or Delayed Rituximab to Eliminate Hairy Cell Leukemia Minimal Residual Disease
Brief Title: Cladribine With Simultaneous or Delayed Rituximab to Treat Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090005; 09-C-0005; NCT00781235 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Hairy Cell Leukemia
Keywords: Hairy Cell Leukemia; Cladribine; Rituximab; Minimal Residual Disease; Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell; Neoplasm, Residual; Leukemia | interventions — Cladribine; Rituximab; Magnetic Resonance Imaging; Electrocardiography; Echocardiography; Caves; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 1/Cladribine with immediate Rituximab (Experimental): Cladribine with immediate Rituximab.
  Interventions: Drug: Cladribine; Drug: Rituximab; Procedure: BMbx; Diagnostic Test: MRI; Diagnostic Test: EKG; Diagnostic Test: Echocardiogram; Diagnostic Test: Abdominal/splenic ultrasound; Procedure: Stress test
- 2/Cladribine with Rituximab Delayed by at Least 6 months After Cladribine (Active Comparator): Cladribine with Rituximab delayed by at least 6 months after Cladribine if and when minimal residual disease is detected.
  Interventions: Drug: Cladribine; Drug: Rituximab; Procedure: BMbx; Diagnostic Test: MRI; Diagnostic Test: EKG; Diagnostic Test: Echocardiogram; Diagnostic Test: Abdominal/splenic ultrasound; Procedure: Stress test
- 3/Non-randomized Group Receiving Cladribine with Immediate Rituximab (Experimental): Non-randomized group receiving Cladribine with immediate Rituximab (before rather than after the 1st of the 5 daily doses of cladribine on day 1).
  Interventions: Drug: Cladribine; Drug: Rituximab; Procedure: BMbx; Diagnostic Test: MRI; Diagnostic Test: EKG; Diagnostic Test: Echocardiogram; Diagnostic Test: Abdominal/splenic ultrasound; Procedure: Stress test

INTERVENTIONS:
Drug: Cladribine — Cladribine 0.15 mg/Kg/day by 2-hour intravenous (i.v.) infusion days 1-5. The infusion time may be changed to 1 hour at the discretion of the principal investigator (PI).
  Other Names: Mavenclad
Drug: Rituximab — Rituximab 375 mg/m^2 intravenous (i.v.) infusion every week x8, begin day 1 in half of randomized patients and in all hairy cell leukemia variant (HCLv) patients, and then again in all patients at least 6 months later when hairy cell leukemia (HCL) is detected by blood fluorescence-activated cell sorting (FACS).
  Other Names: Rituxan
Procedure: BMbx — Baseline and week 5.
  Other Names: Bone marrow biopsy
Diagnostic Test: MRI — Baseline and week 5.
  Other Names: Magnetic resonance imaging
Diagnostic Test: EKG — Baseline and week 5.
  Other Names: Electrocardiogram
Diagnostic Test: Echocardiogram — Baseline.
  Other Names: Echo
Diagnostic Test: Abdominal/splenic ultrasound — Baseline and week 5.
  Other Names: Abdominal/splenic U/S
Procedure: Stress test — Baseline.

SUMMARY:
Background:

Hairy cell leukemia (HCL) is highly responsive to but not curable by cladribine (CdA). HCL responds to rituximab, which is not yet standard therapy for HCL.

Patients with the interleukin 2 (IL-2) receptor (CD25)-negative hairy cell leukemia variant (HCLv) respond poorly to initial cladribine but do respond to rituximab in anecdotal reports.

Deoxycytidine kinase phosphorylates cladribine to chlorodeoxyadenosine triphosphate (CdATP), which incorporates into deoxyribonucleic acid (DNA), leading to DNA strand breaks and inhibition of DNA synthesis. Rituximab is an anti-cluster of differentiation 20 (CD20) monoclonal antibody which induces apoptosis and either complement or antibody dependent cytotoxicity (antibody-dependent cellular cytotoxicity (ADCC) or complement-dependent cytotoxicity (CDC).

Patients in complete remission (CR) to cladribine have minimal residual disease (MRD) by immunohistochemistry of the bone marrow biopsy (BMBx IHC), a risk for early relapse. Tests for HCL MRD in blood or marrow include flow cytometry fluorescence-activated cell sorting (FACS) or polymerase chain reaction (PCR) using consensus primers. The most sensitive HCL MRD test is real-time quantitative PCR using sequence-specific primers real-time quantitative reverse transcriptase polymerase chain reaction (RQ-PCR).

In studies with limited follow-up, MRD detected by tests other than RQ-PCR can be eliminated by rituximab after cladribine in greater than 90 percent of patients, but MRD rates after cladribine alone are unknown. Simultaneous cladribine and rituximab might be superior or inferior to delaying rituximab until detection of MRD.

Only 4 HCL-specific trials are listed on Cancer.gov: a phase II trial of cladribine followed 4 weeks later by 8 weekly doses of rituximab, and phase I-II trials of recombinant immunotoxins targeting cluster of differentiation-22 (CD22) (BL22, HA22) and CD25 (LMB-2).

Objectives:

Primary:

To determine if HCL MRD differs at 6 months after cladribine with or without rituximab administered concurrently with cladribine.

Secondary:

* To compare cladribine plus rituximab vs cladribine alone in terms of 1) initial MRD-free survival and disease-free survival, and 2) response to delayed rituximab for relapse, to determine if early rituximab compromises later response.
* To determine if MRD levels and tumor markers (soluble CD25 and CD22) after cladribine and/or rituximab correlate with response and clinical endpoints.
* To determine, using MRD and tumor marker data, when bone marrow biopsy (BMBx) can be avoided.
* To compare response and MRD after the 1st and 2nd courses of cladribine.
* To evaluate the effects of cladribine and rituximab on normal T- and B-cells.
* To enhance the study of HCL biology by cloning, sequencing and characterizing monoclonal immunoglobulin rearrangements.

Eligibility:

HCL with 0-1 prior courses of cladribine and treatment indicated.

Design:

Cladribine 0.15 mg/Kg/day times 5 doses each by 2hour(hr) intravenous (i.v.) infusion (days 1-5)

Rituximab 375 mg/m^2/week times 8 weeks, randomized half to begin day 1, then repeat for all patients with blood-MRD relapse at least 6 months after cladribine. Also, may repeat for those with blood-MRD relapse at least 6 months after delayed rituximab.

MRD tests used for the primary objective will be limited to BMBx IHC, blood FACS or blood consensus PCR, all Clinical Laboratory Improvement Amendments (CLIA) certified. Blood MRD relapse is defined as FACS positivity or low blood counts (ANC less than 1500/microl, platelet (Plt) less than 100,000/microl, or hemoglobin (Hgb) less than 11).

Stratification: 68 patients with 0 and 62 with 1 prior course of cladribine.

Statistics: 80% power to discriminate rates of MRD of 5 vs 25%, or 10 vs 35%

Non-randomized arm: 20 with HCLv will begin rituximab with cladribine.

Accrual Ceiling: 152 patients (130 HCL, 2 extra HCL if needed, and 20 HCLv.)

DETAILED DESCRIPTION:
Background:

Hairy cell leukemia (HCL) is highly responsive to but not curable by cladribine (CdA). HCL responds to rituximab, which is not yet standard therapy for HCL.

Patients with the interleukin 2 (IL-2) receptor (CD25)-negative hairy cell leukemia variant (HCLv) respond poorly to initial cladribine but do respond to rituximab in anecdotal reports.

Purine analogs cladribine and pentostatin have similar efficacy for HCL, both inhibiting deoxyribonucleic acid (DNA) synthesis selectively in HCL cells. Cladribine is effective after just 1 cycle. Rituximab is an anti-cluster of differentiation 20 (CD20) monoclonal antibody which induces apoptosis and either complement or antibody dependent cytotoxicity (antibody-dependent cellular cytotoxicity (ADCC) or complement-dependent cytotoxicity (CDC).

Patients in complete remission (CR) to cladribine have minimal residual disease (MRD) by immunohistochemistry of the bone marrow biopsy (BMBx IHC), a risk for early relapse. Tests for HCL MRD in blood or marrow include flow cytometry fluorescence-activated cell sorting (FACS) or polymerase chain reaction (PCR) using consensus primers. The most sensitive HCL MRD test is real-time quantitative PCR using sequence-specific primers real-time quantitative reverse transcriptase polymerase chain reaction (RQ-PCR).

In studies with limited follow-up, MRD detected by tests other than RQ-PCR can be eliminated by rituximab after cladribine in > 90% of patients, but MRD rates after purine analog alone are unknown. Simultaneous cladribine and rituximab might be superior or inferior to delaying rituximab until detection of MRD.

Only 4 HCL-specific trials are listed on Cancer.gov: a phase II trial of cladribine followed 4 weeks later by 8 weekly doses of rituximab, and phase I-II trials of recombinant immunotoxins targeting cluster of differentiation-22 (CD22) (BL22, HA22) and CD25 (LMB-2).

Objective:

To determine if HCL MRD differs at 6 months after cladribine with or without rituximab administered concurrently with cladribine.

Eligibility:

HCL with 0-1 prior courses of cladribine or pentostatin and treatment indicated.

Design:

Cladribine 0.15 mg/Kg/day times 5 doses each by 2hour(hr) intravenous (i.v.) infusion (days 1-5)

Rituximab 375 mg/m^2/week times 8 weeks, randomized half to begin day 1, then repeat for all patients with blood-MRD relapse at least 6 months after cladribine. Also, may repeat for those with blood-MRD relapse at least 6 months after delayed rituximab.

MRD tests used for the primary objective will be limited to BMBx IHC, blood FACS, and

bone marrow aspirate FACS, all Clinical Laboratory Improvement Amendments (CLIA) certified. Blood MRD relapse is defined as FACS positivity or low blood counts (absolute neutrophil count (ANC) less than 1500/microl, platelet (Plt) less than 100,000/microl, or hemoglobin (Hgb) less than 11) attributed to HCL. Patients FACS-negative in both blood and bone marrow aspirate are considered MRD-negative complete response (CR) regardless of blood counts.

Randomization: 68 HCL patients with 0 and 62 with 1 prior course of purine analog

Statistics: 80% power to discriminate rates of MRD of 5 vs. 25%, or 10 vs. 35%

Non-randomized HCLv arm: 20 patients with HCLv will begin rituximab with cladribine.

Non-randomized HCL arm: 25 newly diagnosed patients will be enrolled to receive rituximab

beginning day 1, but beginning before the 1st dose of cladribine, rather than after.

Accrual ceiling: 175 evaluable patients (155 HCL and 20 HCLv)

ELIGIBILITY:
* INCLUSION CRITERIA:

Evidence of Hairy Cell Leukemia (HCL) by flow cytometry, reviewed by the Laboratory of Pathology, National Cancer Institute (NCI), including positivity for Cluster of Differentiation 19 (CD19), Cluster of Differentiation 22 (CD22), cluster of differentiation 20 (CD20), and integrin alpha X (CD11c).

Bone marrow biopsy (BMBx) consistent with HCL, reviewed by Laboratory of Pathology, NCI. BMBx may be negative in hairy cell leukemia variant, (HCLv) in patients with increasing peripheral blood HCLv cells and spleen size.

Treatment indicated based on demonstration of at least one of the following, no more than 4 weeks from the time of enrollment, and no less than 6 months after prior purine analog and no less than 4 weeks after other prior treatment, if applicable.

* Neutropenia (absolute neutrophil count (ANC) less than 1000 cells/microl).
* Anemia (hemoglobin (Hgb) less than 10g/dL).
* Thrombocytopenia (Platelet (Plt) less than 100,000/microl).
* Absolute lymphocyte count (ALC) of greater than 5,000 cells/microL
* Symptomatic splenomegaly.
* Enlarging lymph nodes greater than 2cm.
* Repeated infections requiring oral or intravenous (i.v.) antibiotics.
* Patients who have eligible blood counts within 4 weeks from enrollment will not be considered ineligible if subsequent blood counts prior to enrollment fluctuate and become ineligible up until the time of enrollment.

No prior purine analog therapy except up to 1 prior course of cladribine.

No prior rituximab unless HCLv patient.

Eastern Cooperative Oncology Group (ECOG) performance status (78) of 0-3.

Patients must be able to understand and give informed consent.

Women of child-bearing age and all men must use birth control of any type until at least 12 months after the last dose of therapy.

Creatinine less than or equal to 1.5 or creatinine clearance greater than or equal to 60 ml/ml.

Bilirubin less than or equal to 2 unless consistent with Gilbert's (total/direct greater than 5), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 times upper limits of normal.

No other therapy (i.e. chemotherapy, interferon) for 4 weeks prior to study entry, or cladribine for 6 months prior to study entry.

Age at least 18

Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.

Subject has provided written informed consent

Patients must be willing to co-enroll in the investigators companion protocol 10-C-0066 titled Collection of Human Samples to Study Hairy Cell and other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment.

EXCLUSION CRITERIA:

Presence of active untreated infection

Uncontrolled coronary disease or New York Heart Association Classification (NYHA) class III-IV heart disease.

Known infection with HIV. Hepatitis B is allowed only if viral load is undetectable and if on anti-hepatitis B therapy like Entecavir. Hepatitis C is allowed only if viral load is undetectable, and if the patient has received curative therapy.

Patients with documented history of no response to cladribine, and without 50% improvement in platelets, hemoglobin or granulocytes. This exclusion does not apply to HCLv. These patients are eligible regardless of prior response to chlorodeoxyadenosine (CDA)

Pregnant or lactating women.

Presence of active 2nd malignancy requiring treatment. 2nd malignancies with low activity which do not require treatment (i.e. low-grade prostate cancer, basal cell or squamous cell skin cancer) do not constitute exclusions.

Inability to comply with study and/or follow-up procedures.

Presence of central nervous system (CNS) disease, which is symptomatic.

At the Investigators discretion, receipt of a live vaccine within 4 weeks prior to randomization. Efficacy and/or safety of immunization during periods of B-cell depletion have not been adequately studied. It is recommended that a patients vaccination record and possible requirements be reviewed. Per the investigator's discretion, the patient may have any required vaccination/booster administered at least 4 weeks prior to the initiation of study treatment. Review of the patient s immunization status for the following vaccinations is recommended: tetanus; diphtheria; influenza; pneumococcal polysaccharide; Varicella; measles, mumps and rubella (MMR); and hepatitis B. Patients who are considered to be at high risk for hepatitis B virus (HBV) infection and for whom the investigator has determined that immunization is indicated should complete the entire HBV vaccine series at least 4 weeks prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2030-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Bouroncle BA. Thirty-five years in the progress of hairy cell leukemia. Leuk Lymphoma. 1994;14 Suppl 1:1-12. PMID 7820038
- [Background] Kreitman RJ, Cheson BD. Malignancy: Current Clinical Practice: Treatment of Hairy Cell Leukemia at the Close of the 20th Century. Hematology. 1999;4(4):283-303. doi: 10.1080/10245332.1999.11746452. PMID 11399570
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Derived] Chihara D, Arons E, Stetler-Stevenson M, Yuan C, Wang HW, Zhou H, Raffeld M, Xi L, Steinberg SM, Feurtado J, James-Echenique L, Tai CH, Patel KP, Braylan RC, Calvo KR, Maric I, Dulau-Florea A, Kreitman RJ. Long term follow-up of a phase II study of cladribine with concurrent rituximab with hairy cell leukemia variant. Blood Adv. 2021 Dec 14;5(23):4807-4816. doi: 10.1182/bloodadvances.2021005039. PMID 34607348
- [Derived] Chihara D, Arons E, Stetler-Stevenson M, Yuan CM, Wang HW, Zhou H, Raffeld M, Xi L, Steinberg SM, Feurtado J, James L, Wilson W, Braylan RC, Calvo KR, Maric I, Dulau-Florea A, Kreitman RJ. Randomized Phase II Study of First-Line Cladribine With Concurrent or Delayed Rituximab in Patients With Hairy Cell Leukemia. J Clin Oncol. 2020 May 10;38(14):1527-1538. doi: 10.1200/JCO.19.02250. Epub 2020 Feb 28. PMID 32109194
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0005.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab; Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab: Participants with Hairy Cell Leukemia (HCL) with (62 participants) and without (68 participants) prior course of purine analog to be randomized between Arm 1 and Arm 2 (randomization stratified based upon prior purine analog [yes/no]). Cladribine + Rituximab.
- Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected); Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected): Participants with Hairy Cell Leukemia (HCL) with (62 participants) and without (68 participants) prior course of purine analog to be randomized between Arm 1 and Arm 2 (randomization stratified based upon prior purine analog [yes/no]). Cladribine (+ Rituximab after 6 months if minimal residual disease (MRD) detected).
- Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1): Participants with Hairy Cell Leukemia (HCL) without prior course of purine analog to be directly assigned to Arm 3 (25 participants; after completion of the 68 participants without prior purine analog in Cohort 1). Cladribine + Rituximab (Rituximab will be administered just before rather than after the 1st of the 5 daily doses of cladribine
- Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine: Participants with Hairy Cell Leukemia Variant (HCLv) to be directly assigned to Arm 3 (20 participants). Cladribine + Rituximab (Rituximab will be administered just before rather than after the 1st of the 5 daily doses of cladribine
Period: Overall Study
Arm/Group | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine
Started | 34 | 32 | 34 | 30 | 25 | 20
Disease Progression on Study | 1 | 0 | 0 | 0 | 0 | 4
Refused Further Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Death During Follow-up Period | 0 | 0 | 0 | 0 | 0 | 2
Completed | 32 | 28 | 32 | 29 | 25 | 20
Not Completed | 2 | 4 | 2 | 1 | 0 | 0
Not completed — Refused further treatment | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Switched to alternative treatment | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death on study | 2 | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine | Total
Number analyzed (Participants) | 34 | 32 | 34 | 30 | 25 | 20 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 31 | 27 | 19 | 9 | 143
  >=65 years | 5 | 4 | 3 | 3 | 6 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.03 (11.8) | 54.56 (10.23) | 47.94 (11.19) | 51.83 (10.62) | 53.16 (13.85) | 64.7 (11.75) | 53.08 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 5 | 6 | 6 | 5 | 32
  Male | 26 | 30 | 29 | 24 | 19 | 15 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 2 | 0 | 0 | 11
  Not Hispanic or Latino | 0 | 29 | 26 | 28 | 25 | 20 | 128
  Unknown or Not Reported | 32 | 1 | 3 | 0 | 0 | 0 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 1 | 3
  White | 30 | 32 | 30 | 26 | 25 | 18 | 161
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 4 | 1 | 0 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 34 | 30 | 25 | 20 | 175

OUTCOME MEASURES:

1. Primary Outcome: Response Rate Comparing Minimal Residual Disease (MRD) at 6 Months After Start of Treatment in Comparison Groups
Description: Participants with newly diagnosed Hairy Cell Leukemia (HCL) and once relapsed HCL were split and both groups were randomized to receive either simultaneous treatment with Cladribine and Rituxan or Cladribine with Rituxan given no earlier than 6 months after cladribine as needed. Outcome measured by Bone Marrow and Blood Flow cytometry and histochemistry of the core biopsy at the 6 months after start of treatment time point. If all three were negative for hairy cells participants were in a minimal residual disease status (MRD). And were considered without HCL disease at that time point.
Time Frame: Restaged 6 months after the start of treatment
Population: Cohort 2, Arm 3 and Cohort 3, Arm 3 are not reported because the investigator is only comparing the randomized groups. The primary goal is comparing the randomization and Cohort 2 was not randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected)
Number analyzed (Participants) | 34 | 32 | 34 | 30
Percentage of participants | 97.1 | 62.5 | 23.5 | 3.3

2. Secondary Outcome: Minimal Residual Disease (MRD)-Free Survival After Cladribine and up to 2 Courses of Rituximab
Description: Compare Cladribine + Rituxan vs cladribine alone in terms of MRD-free survival. MRD free survival time is the time until relapsing from MRD to -free to Complete response. Measured by blood and bone marrow flow cytometry, complete blood count (CBC), and bone marrow immunohistochemistry.
Time Frame: Testing done 6 months post first dose of treatment, then yearly x2 years and then every 2 years after cladribine indefinitely
Reporting Status: Not Posted, anticipated posting 2030-01

3. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAEv3.0)
Description: Here is the number of participants with serious and/or non-serious adverse events (AE's) assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From first study intervention,Study Day 1, Cycle 1-30 days after study agent up to day 35 for participants receiving cladribine only, up to day 80 for participants receiving cladribine+rituximab, &up to day 80 for participants receiving delayed rituximab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine
Number analyzed (Participants) | 34 | 32 | 34 | 30 | 25 | 20
Participants | 34 | 31 | 34 | 29 | 24 | 19

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed up to 16 years. Adverse Events was monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent, up to day 35 for participants receiving cladribine only, up to day 80 for participants receiving cladribine plus rituximab, and up to day 80 for participants receiving delayed rituximab.
Groups:
- Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab; Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab: Participants with Hairy Cell Leukemia (HCL) with (62 participants) and without (68 participants) prior course of purine analog to be randomized between Arm 1 and Arm 2 (ramdomization stratified based upon prior purine analog [yes/no]). Cladribine + Rituximab.
- Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected); Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected): Participants with Hairy Cell Leukemia (HCL) with (62 participants) and without (68 participants) prior course of purine analog to be randomized between Arm 1 and Arm 2 (ramdomization stratified based upon prior purine analog [yes/no]). Cladribine (+ Rituximab after 6 months if minimal residual disease (MRD) detected).
Arm/Group | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine
All-Cause Mortality (participants affected / at risk) | 2/34 | 2/32 | 0/34 | 1/30 | 0/25 | 5/20
Serious Adverse Events (participants affected / at risk) | 4/34 | 2/32 | 2/34 | 5/30 | 4/25 | 3/20
Other Adverse Events (participants affected / at risk) | 34/34 | 31/32 | 34/34 | 29/30 | 24/25 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab (N=34) | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab (N=32) | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) (N=34) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) (N=30) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) (N=25) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine (N=20)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bladder (urinary)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Arm 1 SubGroup 1 -Cladribine + Rituximab (N=34) | Cohort 1 Arm 1 SubGroup 2 -Cladribine + Rituximab (N=32) | Cohort 1 Arm 2 SubGroup 1-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) (N=34) | Cohort 1 Arm 2 SubGroup 2-Cladribine(+Rituximab After 6 Months if Minimal Residual Disease Detected) (N=30) | Cohort 2 Arm 3 SubGroup 1-Cladribine (Rituximab Before 1st of 5 Daily Doses of Cladribine on Day 1) (N=25) | Cohort 3Arm3 HairyCell LeukemiaVariant-Cladribine +(Rituximab Before 1st of 5 Daily Doses Cladribine (N=20)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 14 (16) | 3 (4) | 9 (10) | 5 (5) | 4 (4) | 3 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 12 (13) | 3 (3) | 10 (11) | 2 (2) | 5 (6) | 6 (6)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 11 (11) | 7 (7) | 10 (13) | 10 (10) | 4 (4) | 6 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 5 (7) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 5 (5) | 5 (7) | 2 (3) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 count (Blood and lymphatic system disorders) | 1 (1) | 3 (7) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 6 (7) | 2 (2) | 1 (1)
Cardiac Arrhythmia - Other (Specify: Sinus Tachycardia) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrhythmia - Other (Specify: Sinus Tachycardia) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrhythmia - Other (Specify: Systolic hypertension) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Specify: Sinus tachycardia) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Constitutional Symptoms - Other (Specify: Joint-effusion) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 6 (7) | 5 (5) | 1 (1) | 4 (5)
Creatinine (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (3) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 19 (21) | 3 (4) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 4 (4)
Edema: limb (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid dysfunction (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5) | 3 (3) | 8 (8) | 4 (5) | 3 (3) | 4 (4)
Febrile neutropenia (Infections and infestations) | 11 (11) | 1 (2) | 8 (8) | 1 (1) | 4 (4) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 14 (14) | 8 (8) | 6 (6) | 6 (7) | 0 (0) | 4 (4)
Fibrinogen (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 12 (12) | 9 (12) | 5 (5) | 9 (11) | 1 (1) | 4 (4)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haptoglobin (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 15 (24) | 14 (21) | 13 (15) | 14 (20) | 12 (25) | 5 (5)
Hemoglobinuria (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hemorrhage, pulmonary/upper respiratory::Larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Specify: Epistaxis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Specify: Macular) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bladder (urinary)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Rectum
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Scrotum
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Sinus
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Wound
Infection - Other (Specify: Pneumonia) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Abdomen NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Muscle (infection myositis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Penis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Spleen (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 24 (39) | 21 (30) | 28 (43) | 17 (22) | 5 (7) | 9 (9)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphatics - Other (Specify: Edema/ankles) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphatics - Other (Specify: Edema: head-and-neck) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 28 (45) | 22 (42) | 29 (44) | 21 (39) | 5 (10) | 14 (18)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 9 (9) | 2 (2) | 2 (2) | 3 (3)
Mood alteration::Anxiety (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 7 (8) | 4 (6) | 2 (2) | 7 (7)
Neurology - Other (Specify: Dizziness) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: cranial::CN II Vision (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: cranial::CN VIII Hearing and balance (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14 (21) | 14 (14) | 19 (25) | 15 (21) | 2 (2) | 5 (5)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (Specify: Extremity-Limb) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify: Extremity-limb, related to BMBx) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Other (Specify: Extremity/Limb) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (Specify: RE limb) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify: with urination) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 6 (6) | 1 (1) | 7 (8) | 2 (2) | 2 (2) | 3 (3)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Cardiac/heart (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Pain::Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain::Face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 11 (11) | 7 (8) | 11 (12) | 4 (5) | 3 (4) | 3 (3)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (5) | 3 (3) | 2 (3) | 1 (1) | 4 (4)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain::Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Scrotum (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pain::Urethra (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 13 (15) | 9 (10) | 5 (8) | 7 (8) | 4 (6) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 24 (29) | 17 (24) | 6 (11) | 7 (12) | 6 (8) | 9 (9)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4) | 8 (8) | 3 (3) | 1 (1) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 14 (15) | 4 (4) | 16 (16) | 4 (4) | 3 (5) | 6 (6)
Rash: dermatitis associated with radiation::Chemoradiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify: Hyperuricemia) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 17 (19) | 9 (9) | 9 (11) | 4 (4) | 9 (10) | 8 (8)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular arrhythmia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0) | 6 (7) | 5 (5) | 2 (2) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia::Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT00923013/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Eligibility Screening Consent (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT00923013/ICF_001.pdf
  • Informed Consent Form: Cohort Non-Randomized, Classic Hairy Cell Consent (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT00923013/ICF_002.pdf
  • Informed Consent Form: Cohort Non-Randomized Consent (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT00923013/ICF_003.pdf
  • Informed Consent Form: Cohort Randomized Consent (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT00923013/ICF_004.pdf